CLINICAL TRIAL: NCT03885440
Title: Age and Sleep Apnea Syndrome: Clinical Features and Outcomes
Brief Title: Age and Sleep Apnea Syndrome
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Taipei Veterans General Hospital, Taiwan (Other Government)
Responsible Party: Principal Investigator, vghtpe user, Principal Investigator, Medical Doctor, Taipei Veterans General Hospital, Taiwan
Other Study IDs: 2018-10-002CC
Record Dates: First submitted 2019-03-16; First posted 2019-03-21 (Actual); Last update posted 2019-04-09 (Actual); Status verified 2019-04

CONDITIONS: OSA; Age Problem
MeSH Terms: interventions — Aging

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (4):
- Young adult, without OSAS: 20<=Age<40 years old, apnea-hypopnea index(AHI)<5
  Interventions: Other: Age
- Young adult, with OSAS: 20<=Age<40 years old, AHI>=5
  Interventions: Other: Age; Other: OSA
- older adult, without OSAS: Age>=40 years old, AHI<5
- older adult, with OSAS: Age>=40 years old, AHI>=5
  Interventions: Other: OSA

INTERVENTIONS:
Other: Age — Age<40 years old is chosen as the cutoff value.
  Groups: Young adult, with OSAS; Young adult, without OSAS
Other: OSA — The diagnosis of OSA (obstructive sleep apnea) relies on polysomnographic data showing an apnea-hypopnea index at least 5/hr with compatible symptoms.
  Groups: Young adult, with OSAS; older adult, with OSAS

SUMMARY:
By clinical record review, this retrospective study aims to compare the different age groups of patients with obstructive sleep apnea, who were diagnosed and treated in Taipei Veterans General Hospital, Taiwan.

DETAILED DESCRIPTION:
This retrospective study aims to compare the characteristics of patients with obstructive sleep apnea (OSA). Patients with sleep problem and received a prior polysomnography at Taipei Veterans General Hospital during Jan. 1, 2016 to Dec. 31, 2017 will be enrolled. Obstructive sleep apnea (OSA) is defined by an apnea-hypopnea index(AHI) at least 5/hr with compatible symptoms. Their clinical record will be reviewed and data including demography, polysomnography, comorbidities and details related to upper airway structure will be collected. The charactereistics would be compared with Student's t tests, Mann-Whitney U tests, or Chi square tests if appropriated.

ELIGIBILITY:
Inclusion Criteria:

* Patients with sleep complaints and received PSG in sleep center in Taipei Veterans General Hospital

Exclusion Criteria:

* Patients who ever received treatment for OSA
* Patients cannot tolerate PSG examination
* Patients cannot complete the questionnaires before and after PSG examination

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adults with sleep complaints
Sampling Method: Non-Probability Sample
Enrollment: 3000 (Estimated)
Dates: Start 2019-04-08 (Actual); Primary Completion 2019-06-30 (Estimated); Study Completion 2019-09-30 (Estimated)

PRIMARY OUTCOMES:
Apnea-hypopnea index(AHI) | through study completion, an average of 1 year
  Counts of apnea/hypopnea events per hour

SECONDARY OUTCOMES:
Body mass index(BMI) | through study completion, an average of 1 year
  The body mass divided by the square of the body height.
Posterior airway space (PAS) | through study completion, an average of 1 year
  The diameter from supramentale to gonion.
Number of participants with comorbidities | through study completion, an average of 1 year
  Self-reported comorbidities including cardiovascular disease, stroke, hypertension, diabetes mellitus, hyperlipidemia, lung disease, anxiety, depression.
Sleep efficiency | through study completion, an average of 1 year
  The ratio of the total time spent asleep (total sleep time) in a night compared to the total amount of time spent in bed.
arousal index | through study completion, an average of 1 year
  The number of arousals and awakenings as a frequency per hour of sleep.
oxygen desaturation index | through study completion, an average of 1 year
  The number of times per hour of sleep that the blood's oxygen level drop by 4% from baseline.

CONTACTS AND LOCATIONS:
Locations (1):
- Chest department, Taipei Veteran General Hospital, Taipei, Taiwan

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Chiu HY, Chou KT, Su KC, Lin FC, Liu YY, Shiao TH, Chen YM. Obstructive sleep apnea in young Asian adults with sleep-related complaints. Sci Rep. 2022 Nov 29;12(1):20582. doi: 10.1038/s41598-022-25183-5. PMID 36447027